CLINICAL TRIAL: NCT03212066
Title: Elementary School Mindfulness-Based Substance Use Prevention Program
Brief Title: Master Mind Program Evaluation Study
Acronym: MasterMind
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Innovation Research & Training (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R44AA021342 (NIH); R44AA021342 (NIH)
Record Dates: First submitted 2017-07-05; First posted 2017-07-11 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Substance Abuse; Mindfulness
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Master Mind is a 25-lesson elementary school, mindfulness education substance abuse prevention program for 4th and 5th grade classrooms.
  Interventions: Behavioral: Master Mind
- Wait-List Control (No Intervention): Business as usual

INTERVENTIONS:
Behavioral: Master Mind — Master Mind is a 25-lesson elementary school mindfulness education substance abuse prevention program. Each lesson takes approximately 15 minutes and is designed to be taught by trained teachers every day for 5 weeks.
  Arms: Intervention

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial to evaluate the efficacy of the Master Mind program, a mindfulness education substance abuse prevention program. The program has the goal of enhancing coping strategies and decision-making skills and preventing substance abuse in late elementary school students.

ELIGIBILITY:
Inclusion Criteria:

* English Fluency

Exclusion Criteria:

-

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 518 (Actual)
Dates: Start 2017-08-23 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Change in score on Positive and Negative Affect Scale for Children - Shortened Version (PANAS) | 6 weeks
  Assesses students' experiences of positive and negative emotions.
Change in score on Self-Report Coping Measure | 6 weeks
  Assesses students' coping in response to stressors.
Change in score on Intentions to use alcohol or tobacco | 6 weeks
  Assesses students' intentions to use alcohol or tobacco in the future.
Change in score on Willingness to use alcohol or tobacco | 6 weeks
  Assesses students' willingness to use alcohol or tobacco by responding to imagined situations.
Change in score on The Peer Relations questionnaire | 6 weeks
  Assesses students' feelings about their classmates.
Change in score on The Emotional Self-Efficacy Scale for Youth | 6 weeks
  Assesses students' beliefs about their ability to manage emotions.
Change in scores on Flanker Inhibitory Control and Attention Test | 6 weeks
  Assesses students' executive functioning skills via a performance task.
Change in score on Childhood Executive Functioning Inventory (CHEXI) | 6 weeks
  Assesses teacher ratings of students' executive functioning.
Change in score on The Child Behavior Scale (CBS) | 6 weeks
  Assesses teacher ratings of student behavior and peer relationships.
Change in Iowa Conners Teacher Rating Scale | 6 weeks
  Assesses teacher ratings of students' inattention and aggression.
Change in Iowa Conners Teacher Rating Scale | 14 weeks
  Assesses teacher ratings of students' inattention and aggression.
Change in Student grades | 6 weeks
  Teachers will be asked to provide grades for each student for Math and Language Arts.
Change in Student grades | 14 weeks
  Teachers will be asked to provide grades for each student for Math and Language Arts.

SECONDARY OUTCOMES:
Student Consumer Satisfaction Questionnaire | 6 weeks
  Assesses the overall opinions of students in the intervention group about the Master Mind lessons and activities.
Teacher Program Feasibility Questionnaire | 6 weeks
  Assesses the overall opinions of teachers in the intervention group related to feasibility of the Master Mind program.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Parker, PhD, Principal Investigator — Innovation Research & Training
Locations (1):
- innovation Research & Training, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Parker AE, Kupersmidt JB, Mathis ET, Scull TM, Sims C. The impact of mindfulness education on elementary school students: Evaluation of the Master Mind Program. Adv Sch Ment Health Promot. 2014;7(3):184-204. doi: 10.1080/1754730X.2014.916497. Epub 2014 May 19. PMID 27057208